CLINICAL TRIAL: NCT04287010
Title: The Effect of Intra-dialytic Potassium and Magnesium Fluctuations on Cardiovascular Functioning in ESRD Patients Undergoing In Center Hemodialysis
Brief Title: Potassium Flux in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Frank O'Brien, Assistant Professor of Medicine. Nephrology, Washington University School of Medicine
Other Study IDs: 201901179
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current practice of outpatient hemodialysis entails prescription of standard electrolyte concentrations based upon patient prescription history and monthly serum electrolyte measurements. Dialysate concentration of potassium can be adjusted based on standard available concentrations including 2mmol/L and 3mmol/L. Standard available dialysate concentration of Magnesium is 0.5mmol/L (which is not ordinarily adjusted further). Potassium and Magnesium are not routinely measured before or after each dialysis, therefore serum levels are largely unknown outside of once monthly measurements.

This study aims to further study this correlation of electrolyte fluctuations (potassium and magnesium) and cardiac arrhythmias/heart rate variability in the ESRD population.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional study utilizing a study population at Chromalloy American Kidney Center, an outpatient dialysis unit, which currently serves approximately 150 End Stage Renal Disease (ESRD) patients.

After enrollment, patients will be provided with a schedule for data collection. A standard 12-lead ECG will be performed.A small non-invasive device (MyPatch Holter monitor) will be attached to each patient's chest before their first weekly dialysis session to measure heart rhythm and arrhythmia generation. After the recorder is attached, a standard set of bedside autonomic function tests will be administered. These tests include standing from supine position, hand grip, Valsalva maneuver and deep breathing.Changes in heart rate, heart rhythm, and blood pressure in response to these maneuvers will be assessed. The holter monitor will be worn for the next 92-96 hours and removed after completion of their regular third weekly dialysis session (Friday or Saturday). The data from these holter monitors will be analyzed by the Heart Rate Variability Lab at Washington Univeristy. No modifications to the Holter monitor devices will be made for this study.

Patient vital signs pre/intra/post dialysis by standard protocol will be obtained, including the following parameters: blood pressure, heart rate, oxygen saturation, relative blood volume/hematocrit, dialysate flow rate, blood flow rate, ultrafiltration volume.Participant serum sodium, chloride, potassium, blood urea nitrogen, and magnesium immediately prior to and after dialysis session will be measured. Participant serum potassium and magnesium levels every 30 minutes for the first 2 hours of the first weekly dialysis session will be measured by taking 1mL of blood from the dialysis circuit. Effluent dialysate, which contains no blood or cellular components, will be collected concurrently with serum sample analysis every 30 minutes during the first weekly dialysis session by taking 10mL of fluid from the dialysate drain line to be analyzed for sodium, chloride, and potassium. Serum potassium levels will also be measured immediately prior to and after second and third weekly dialysis sessions by taking 1mL of blood from dialysis circuit. The capability to draw blood from the dialysis circuit/tubing has already been incorporated as an industry standard and no modifications to standard dialysis circuit will be made. This will ensure that the patient will not have any needle sticks to obtain necessary samples. Obtained serum samples will subsequently be coded and sent to the Core Lab for Clinical Studies (CLCS) at Washington University for processing and destruction there after.

All specimens will be assigned a de-identified study code that will be stored in a secure/locked location separate from collected data. All clinical data obtained will be de-identified and entered into a datasheet on a Washington University secure encrypted server. In addition, the Washington University in St. Louis School of Medicine Institute for Informatics, Informatics Core Services (ICS) will be used for centralized management and processing of collected data. Washington University in St. Louis belongs to a consortium of institutional partners that work to maintain a software toolset and workflow for electronic collection and management of research and clinical trial data. The Research Electronic Data Capture (REDCap) system will be utilized for data collection and processing in our study. The REDCap servers are securely housed in an on-site limited access data center managed by the Research Infrastructure Services at Washington University. All web-based information and transmission are encrypted with storage on a private, firewall protected network.

Data collected by Holter monitors and serum electrolyte measurements will subsequently be analyzed by the research team.

Participation in this study will not interfere with regularly scheduled thrice weekly dialysis treatments and clinic workflow. Nor will participation in this study result in modification of previously prescribed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Consistent thrice weekly in center hemodialysis as defined as no missed sessions in the last 30 days.
* Goal Kt/V Urea (>1.2, which suggests adequate dialysis based on KDOQI guidelines) for at least 3 months
* Serum potassium 3.5-8.0 mEq/L
* Hemoglobin of >8.0g/dL

Exclusion Criteria:

* Age <18 years
* Evidence of residual renal function as defined by >100mL of urine output per day
* Those whom do not have capacity to consent
* Change in dialysis prescription within the past 30 days
* 12-lead ECG shows non-sinus cardiac rhythm (atrial fibrillation, atrial flutter, or paced rhythm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients based on a limited chart review from the Chromalloy American Kidney Center population will be recruited. These will all be on in center hemodialysis three times per week. Eligible patients based on inclusion/exclusion criteria as listed above will be randomly selected by a random number generator. If selected, they will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
To examine and better define the correlation between electrolyte fluctuations, arrhythmia generation, and heart rate variability contributing to cardiovascular morbidity/mortality as described in previous retrospective observational studies. | 1 year
  This study aims to assess if there is a correlation between serum electrolyte changes and abnormal heart rhythms or heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Univeristy in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No sharing planned